CLINICAL TRIAL: NCT02683057
Title: Influence of Physical Exercise on Semen Quality
Status: Completed | Type: Observational
Sponsor: IVI Bilbao (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 1411-BIO-080-RM
Record Dates: First submitted 2016-01-25; First posted 2016-02-17 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Sexual Abstinence
MeSH Terms: conditions — Sexual Abstinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- IPAQ HIgh: Excessive physical activity:IPAQ quantifying the activity physical according vigorous intensity activities at least 3 days per week adding a minimum total physical activity of at least 1500MET-minutes / week or 7 or more days any combination of walking, moderate intensity or vigorous intensity activities a total minimum of physical activity of at least 3,000 MET-minutes / week
  Interventions: Other: International Physical Activity Questionnaire (IPAQ)
- IPAQ Moderate: Ideal Physical activity: IPAQ quantifying the activity physical according 3 days or more of vigorous intensity physical activity at least 20 minutes per day or 5 or more days of moderate intensity and / or walk at least 30 minutes per day or 5 or more days of any combination of walking, moderate-intensity activity and activity vigorous intensity for a total minimum of physical activity of at least 600 MET-minutes / week.
  Interventions: Other: International Physical Activity Questionnaire (IPAQ)
- IPAQ Low: IPAQ quantifying the activity physical according Insufficient physical activity: Individuals who can not put on the criteria of the above categories.
  Interventions: Other: International Physical Activity Questionnaire (IPAQ)

INTERVENTIONS:
Other: International Physical Activity Questionnaire (IPAQ) — all candidates for sperm donors clinic IVI IVI Bilbao and Valencia were will provide the international physical activity questionnaire (IPAQ) attached to analyze the total physical activity. This will be self-completed questionnaire beforeSperm donation. (Appendix 1) Age, snuff, weight, BMI, alcohol, drug use and the type of sport that practices will be analyzed: Additionally a tab for each donor collecting the existence of associated factors be drawn. (Appendix 2)

SUMMARY:
Our study addresses a previously selected population or by physical activity but not for semen quality semen donor candidates donation program within the clinic.

Total physical activity was analyzed according to the universally accepted international physical activity questionnaire (IPAQ) The existence of confounding factors associated She purge age, snuff, weight, BMI, alcohol, drugs, type of sport and associated blood parameters determinations will be made to exercise.

DETAILED DESCRIPTION:
The level of physical activity recommended great unknown and its influence from the therapeutic point of view to improve semen quality.

For it will be held:

* 3 groups of physical activity are established, according to their score in the IPAQ: High, minimum of physical activity between > 1500 MET week Moderate: minimum of physical activity of between 600- 1500 MET week Low : until < 600 MET week
* Implementation of a double analysis: Seminal and hormonal
* Standardization of confounding factors associated with the individual

ELIGIBILITY:
Inclusion Criteria:

* Appear as sperm donor
* Age between 18-35 years
* First sperm donation
* Sexual abstinence 3-5 days
* Having signed informed consent

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Candidates for sperm donors in the donation program which aims clinic It is performed in 432 cases. For that, our study addresses a population previously selected either by physical activity or by semen quality
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Ascertain the influence of physical activity in sperm quality to candidates for sperm donors in the donation program according to the universally accepted questionnaire International physical activity (IPAQ) | 2 years
  Semen parameters will be evaluated according to WHO criteria blinded on clinical and data analyst.
  International Physical Activity Questionnaire (IPAQ) offers before sperm donation quantifying the activity "walk", "activities of moderate intensity" and "vigorous intensity activities" assigned to each activity about energy requirements defined in METs, being multiples of the rate of metabolic rate equivalent to kilocalories for a 60 kg.
  The median and interquartile range (between Q1 and Q3) is calculated for walking (W), activities of moderate intensity (M), activities of vigorous intensity (V) and a combined result of total physical activity. All results must be expressed as continuous METminutos / week.

SECONDARY OUTCOMES:
Existence of confounding factors associated with physical activity | 2 years
  The existence of confounding factors such as age, tobacco, weight, BMI, alcohol, drugs, type of sport will be cleaned and blood parameters associated with physical activity will be defined.
  A data tab/sheet for each donor was made . The existence of related factors such as age, tobacco, weight, BMI, alcohol, drug and the type of sport exercised were been analysed.
  It categorizes the population into quartiles depending on their activity and determine which is which is associated with a better seminal quality the same debugging is made confounding previously mentioned.
  multivariate analysis to determine the correlation between physical activity and sperm parameters

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Matorras, Principal Investigator — IVI Bilbao
Locations (1):
- IVI Bilbao, Leioa, Vizcaya, Spain